CLINICAL TRIAL: NCT05174078
Title: Food as Medicine: A Quasi-Randomized Control Trial of Healthy Foods for Chronic Disease Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cleveland Clinic Akron General (Other)
Collaborators: The Cleveland Clinic (Other); The University of Akron (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21029
Record Dates: First submitted 2021-12-01; First posted 2021-12-30 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Obesity; Hypertension; Pre-diabetes; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Hypertension; Glucose Intolerance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: A quasi-randomized control trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Medically-Tailored Meals (MTM) (Experimental): Medically-tailored meals delivered to participants' homes for 15 weeks AND one medical nutrition therapy session with a dietician + viewership of 2 to 4 nutrition education videos.
  Interventions: Other: Medically-tailored meals
- Produce Box and Recipes (Experimental): Weekly produce box delivered to participants' homes and access to recipes via the internet for 15 weeks AND one medical nutrition therapy session with a dietician + viewership of 2 to 4 nutrition education videos.
  Interventions: Other: Produce box and recipes
- Standard of Care (No Intervention): Matched controls from the same base population as participants in the intervention arms. Controls will identified from the electronic medical record (EMR).

INTERVENTIONS:
Other: Medically-tailored meals — Medically tailored meals delivered to patients' homes for 15 weeks AND one medical nutrition therapy session with a dietician + viewership of 2 to 4 nutrition education videos.
  Arms: Medically-Tailored Meals (MTM)
Other: Produce box and recipes — Weekly produce box and access to recipes via internet for 15 weeks AND one medical nutrition therapy session with a dietician + viewership of 2 to 4 nutrition education videos.
  Arms: Produce Box and Recipes

SUMMARY:
The purpose of this study is to investigate the effect of providing healthy foods and nutrition education on participants' body weight, blood pressure, and average blood sugar level.

The healthy food offerings tested in this study will help determine which option is best to improve health outcomes among Cleveland Clinic Akron General patients with chronic conditions. Findings from this study could guide doctors in deciding on appropriate nutrition and dietitian services for Cleveland Clinic patients.

DETAILED DESCRIPTION:
Participants will receive healthy food items for 15 weeks and nutrition counseling and education to support chronic disease management at no cost. The healthy food items will consist of either medically-tailored pre-prepared meals, or a weekly produce box with recipes depending on the study arm. Participants must complete a baseline study visit, one nutritional counseling session via phone, 2 to 4 nutrition education videos, and a 16-week post-intervention study visit.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older who are patients at Akron General Center for Family Medicine
* Have body mass index (BMI) equal to or greater that 30kg/m2 AND
* Have at least one of the following diagnoses determined based on patients' problem list in the electronic medical record (EMR) and the international classification of diseases, 10th revision (ICD-10) codes:

  1. Pre-type 2 diabetes mellitus
  2. Type 2 diabetes mellitus
  3. Hypertension
* Have NOT participated in nutrition counseling at the University of Akron Nutrition Center within the past 6 months

Exclusion Criteria:

* Food allergies
* Pregnant
* No access to internet
* Need English language interpretation
* Currently participating in a structured weight loss program or using weight loss medications
* Any condition that, in the Investigator's judgement, interferes with the ability to adhere to study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Change in participants' body weight | From baseline visit (W1) to 16 week visit and at 6 months and 12 months from baseline
  Percent weight loss

SECONDARY OUTCOMES:
Pre-type 2 diabetes mellitus: Change in number of medications | From baseline visit (W1) to 16 week visit and at 6 months and 12 months from baseline
  Absolute change in number of medications
Pre-type 2 diabetes mellitus: Change in medication dosage | From baseline visit (W1) to 16 week visit and at 6 months and 12 months from baseline
  Percent change in medication dosage
Pre-type 2 diabetes mellitus: Change in HbA1c | From baseline visit (W1) to 16 week visit and at 6 months and 12 months from baseline
  Absolute change in HbA1c
Type 2 diabetes mellitus: Change in number of medications | From baseline visit (W1) to 16 week visit and at 6 months and 12 months from baseline
  Absolute change in number of medications
Type 2 diabetes mellitus: Change in medication dosage | From baseline visit (W1) to 16 week visit and at 6 months and 12 months from baseline
  Percent change in medication dosage
Type 2 diabetes mellitus: Change in HbA1c | From baseline visit (W1) to 16 week visit and at 6 months and 12 months from baseline
  Absolute change in HbA1c
Hypertension: Change in number of medications | Baseline visit (W1) to 16 week visit
  Absolute change in number of medications
Hypertension: Change in medication dosage | Baseline visit (W1) to 16 week visit
  Percent change in medication dosage
Receipt of healthy food items: The Hunger Vital Sign scale | Baseline visit (W1) to week 16 visit
  Values on the scale are: often true, sometimes true, and never true. A positive response to either or both of the first two values (often true, sometimes true) identifies households as being at risk for food insecurity
Receipt of healthy food items: Eating at America's Table scale | Baseline visit (W1) to week 16 visit
  Each reported frequency is expressed as a daily average ranging from 0 to 5. The estimate of the daily number of Pyramid/MyPyramid servings is calculated as average daily frequency x the number of Pyramid/MyPyramid servings for the portion size, summed across all food groups. A higher score for fruits and vegetables indicates a better outcome.
Receipt of healthy food items: Patient Health Questionnaire-8 Depression Scale | Baseline visit (W1) to week 16 visit
  Eight items, each of which is scored 0 to 3, providing a 0 to 24 severity score. Overall score is the sum of the 8 items. A score of 10 or greater is considered major depression, 20 or more is severe major depression.
Nutrition Education: Healthy Eating and Weight Self-Efficacy Scale | Baseline visit (W1) to 16-week visit
  Values on the scale are: Strongly disagree, disagree, neutral, agree, and strongly agree. Responses of agree and strongly agree indicate a better outcome.
Nutrition Education: Self-Efficacy for Managing Chronic Diseases Scale | Baseline visit (W1) to 16-week visit
  Six items, each of which is scored 0 to 10. Overall score is the mean of the 6 items. A higher score indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Elliot B Davidson, MD, FAAFP, Principal Investigator — Cleveland Clinic Akron General
Locations (1):
- Cleveland Clinic Akron General, Akron, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kibera PW, Ofei-Tenkorang NA, Mullen C, Lear AM, Davidson EB. Food as medicine: a quasi-randomized control trial of two healthy food interventions for chronic disease management among ambulatory patients at an urban academic center. Prim Health Care Res Dev. 2023 Dec 21;24:e72. doi: 10.1017/S1463423623000579. PMID 38126528